CLINICAL TRIAL: NCT03483220
Title: Relation Between Emotional Regulation and Impulsivity in Cannabis Use Disorder and the Morphometric Changes in Brain Reward System Structures
Brief Title: Emotional Regulation, Impulsivity in Cannabis Its Relation to MRI Brain Structure
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Mostafa, Lecturer of psychiatry, Assiut University
Other Study IDs: MRI brain study in addiction
Record Dates: First submitted 2018-03-20; First posted 2018-03-30 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Addiction
Keywords: Addiction, MRI, emotional regulation
MeSH Terms: conditions — Behavior, Addictive; Emotional Regulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cases: patients with cannabis use disorder
  Interventions: Diagnostic Test: MRI brain

INTERVENTIONS:
Diagnostic Test: MRI brain — 1. Emotion Regulation Questionnaire (ERQ): A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale .
  UPPS-P Impulsive Behavior Scale- Short form: The UPPS-P impulsivity scale is a 20-item scale designed to assess five distinct personality traits to impulsive behavior: Negative Urgency, Lack of Perseverance, Lack of Premeditation, Positive Urgency and Sensation Seeking .
  Magnetic resonance imaging examination:
  The MR examination of brain was done using 1.5T MR scanner (Achieva, Philips Medical Systems, The Netherlands) with a 16 channel head coil without using any sedation.
  Other Names: Emotion Regulation Questionnaire (ERQ); UPPS-P Impulsive Behavior Scale; structured clinical interview

SUMMARY:
cannabis addiction is a major health hazard that has its effect on personality and behavior including the impulsivity and emotional regulation. It also has its effect on both the structure and function of different brain regions involved in brain reward system.

the aim of the study is to study the emotional regulation and impulsivity among people with cannabis addiction studying the change in the volume of brain reward system structures' volume in relation to cannabis addiction and the change in the mentioned behavioral traits.

DETAILED DESCRIPTION:
Introduction:

Cannabis sativa is a widely used drug comprising a broad spectrum of usage ranging from recreational users to chronic addicts.

Dependence on cannabis is considered a major global health related issue. Cannabis is still considered the most used psychoactive substance worldwide with an estimated 2.8-5.1 % of global adult population has used cannabis in 2019.

Epidemiological studies show that cannabis is the leading drug of abuse in Egypt and in Upper Egypt. Prevalence of cannabis dependence is estimated to be 7.4% in Egypt and 6.66 % in Upper Egypt.

Cannabis dependence is associated with multiple neurobehavioral abnormalities which can be considered as a psychological determinants of cannabis dependence .

There is an increasing evidence of association between emotional dysregulation and dependence on different substances of abuse. Such dysregulation affects both components of emotional regulation; reappraisal and suppression of emotions' expression. The pattern of this dysregulation differs according to the type of substance of dependence and can affect the pattern of substance abuse.

Impulsivity is a proposed endophenotype for substance dependence as well as a possible consequence of prolonged drug use. Drugs of addiction and subconscious craving are likely to increase impulsiveness due to the loss of frontal cortical inhibition of impulses and increased limbic drive. Cannabis use may lead to a loss of attention, reflection and inhibitory control.

Materials and Methods:

This cross-sectional study ran between at the addiction management unit, Assiut University, Egypt. Two groups of participants were recruited in the study: Group (A): 32 patients with cannabis used disorder diagnosed according to DSM-5 criteria recruited from the addiction outpatient clinic at the Hospital of Neurology and Psychiatry at Assiut University. Group (B): 34 healthy individuals as a cross matching control group.

Inclusion criteria were age above 18 years, current chronic cannabis dependence. Exclusion criteria were being in withdrawal state, other psychiatric disorders, and history or current neurological or medical disease.

Ethical considerations:

A signed, informed consent was obtained from patients and their families or caregivers to participate in the study. Confidentiality was maintained during the whole study.

Assessment tools:

All participants were first assessed through a semi-structured interview using the Structured clinical interviews for axis I diagnosis (SCID-I) to rule out any psychiatric comorbidities.

Emotion Regulation Questionnaire (ERQ): A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale.

UPPS-P Impulsive Behavior Scale- Short form: The UPPS-P impulsivity scale is a 20-item scale designed to assess five distinct personality traits to impulsive behavior: Negative Urgency, Lack of Perseverance, Lack of Premeditation, Positive Urgency and Sensation Seeking.

Magnetic resonance imaging examination:

The MR examination of brain was done using 1.5T MR scanner (Achieva, Philips Medical Systems, The Netherlands) with a 16 channel head coil without using any sedation.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Clearly consenting to participate in the study. . patient with substance use disorder

Exclusion Criteria:

* Intoxication or withdrawal state.
* Comorbid Axis I psychiatric disorder.
* any current or past neurological disorder.

Ages: 18 Years to 45 Years | Sex: Male
Age Groups: Adult
Study Population: 66 participants with cannabis use disorder diagnosed by DSM-5 criteria were recruited from addiction unit at Assiut University hospitals
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
degree of impulsivity in addicts | 7 months
  the UPPS-P scale was used to measure the degree of impulsivity. it is a 20-item scale designed to assess five distinct personality traits to impulsive behavior: Negative Urgency, Lack of Perseverance, Lack of Premeditation, Positive Urgency and Sensation Seeking
measuring the volume of prefrontal cortex in addicts | 7 months
  MRI brain with voxel based morphometry was used in measuring the volume of different brain regions involved in the brain reward system

CONTACTS AND LOCATIONS:
Overall Officials: Khaled AM Elbeh, professor, Study Chair — Assiut University; Yasser M Elsorogy, professor, Study Director — Assiut University; Gilan K Ramadan, Lecturer, Study Director — Assiut University; Gehan S Seif, professor, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engel A, Caceda R. Can Decision Making Research Provide a Better Understanding of Chemical and Behavioral Addictions? Curr Drug Abuse Rev. 2015;8(2):75-85. doi: 10.2174/1874473708666150916113131. PMID 26373849
- [Background] Schultz W, Preuschoff K, Camerer C, Hsu M, Fiorillo CD, Tobler PN, Bossaerts P. Explicit neural signals reflecting reward uncertainty. Philos Trans R Soc Lond B Biol Sci. 2008 Dec 12;363(1511):3801-11. doi: 10.1098/rstb.2008.0152. PMID 18829433
- [Background] Nestler EJ, Carlezon WA Jr. The mesolimbic dopamine reward circuit in depression. Biol Psychiatry. 2006 Jun 15;59(12):1151-9. doi: 10.1016/j.biopsych.2005.09.018. Epub 2006 Mar 29. PMID 16566899
- [Background] Cyders MA, Littlefield AK, Coffey S, Karyadi KA. Examination of a short English version of the UPPS-P Impulsive Behavior Scale. Addict Behav. 2014 Sep;39(9):1372-6. doi: 10.1016/j.addbeh.2014.02.013. Epub 2014 Mar 3. PMID 24636739
- [Background] Mohajerin B, Dolatshahi B, Pour Shahbaz A, Farhoudian A. Differences between expressive suppression and cognitive reappraisal in opioids and stimulant dependent patients. Int J High Risk Behav Addict. 2013 Jun;2(1):8-14. doi: 10.5812/ijhrba.8514. Epub 2013 Jun 26. PMID 24971265
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Jakubczyk A, Trucco EM, Kopera M, Kobylinski P, Suszek H, Fudalej S, Brower KJ, Wojnar M. The association between impulsivity, emotion regulation, and symptoms of alcohol use disorder. J Subst Abuse Treat. 2018 Aug;91:49-56. doi: 10.1016/j.jsat.2018.05.004. Epub 2018 May 31. PMID 29910014
- [Background] Gillespie NA, Neale MC, Bates TC, Eyler LT, Fennema-Notestine C, Vassileva J, Lyons MJ, Prom-Wormley EC, McMahon KL, Thompson PM, de Zubicaray G, Hickie IB, McGrath JJ, Strike LT, Renteria ME, Panizzon MS, Martin NG, Franz CE, Kremen WS, Wright MJ. Testing associations between cannabis use and subcortical volumes in two large population-based samples. Addiction. 2018 Apr 24:10.1111/add.14252. doi: 10.1111/add.14252. Online ahead of print. PMID 29691937